CLINICAL TRIAL: NCT03932812
Title: Building a Bridge (Between Clinical and Community Care): Post-diagnosis Support for Persons With Dementia and Their Families
Brief Title: Building a Bridge (BAB) Between Clinical and Community Care
Acronym: BAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sato Ashida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Kansas (Other); University of Michigan (Other); Boston College (Other); Drexel University (Other)
Responsible Party: Sponsor-Investigator, Sato Ashida, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201804835; 1R21AG056716-01A1 (NIH)
Record Dates: First submitted 2019-04-16; First posted 2019-05-01 (Actual); Results first posted 2022-12-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2022-11

CONDITIONS: Caregiver Burden
Keywords: Alzheimer's disease; Dementia; Caregiver; Bridging community; Bridging medical settings
MeSH Terms: conditions — Caregiver Burden; Alzheimer Disease; Dementia | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Options Counselor Health Educator Intervention Group (Experimental): These individuals will receive the Options Counselor Health Educator Intervention
  Interventions: Behavioral: Options Counselor Health Educator (OC-HE) Intervention
- Control (No Intervention): These individuals will receive the typical standard of care treatment from clinics

INTERVENTIONS:
Behavioral: Options Counselor Health Educator (OC-HE) Intervention — The OC-HE will meet in person with the participant one time and five times via telephone to provide options counseling based on modules developed by the research team
  Arms: Options Counselor Health Educator Intervention Group

SUMMARY:
Dementia diagnosis triggers a transitional phase for the individuals and their families, often causing emotional distress and family conflicts due to the ambiguity of the illness and future trajectories. Families often report a lack of information and guidance during the period immediately following diagnosis, suggesting a missed opportunity for prevention of family distress at the outset of the caregiver and patient career. With large and increasing numbers of individuals newly diagnosed with Alzheimer's Disease and Related Dementias (ADRD) each year, there is an urgent need to develop effective intervention models to support role transitions and minimize distress related to ADRD diagnosis. The long-term goal of this research is to minimize negative consequences of ADRD by enhancing the support systems of the affected families as they start their new and challenging phase of life as patients and family caregivers. The aim of this research is to evaluate the impact of this new Options Counselor-Health Education (OC-HE) intervention on bridging the medical and community-settings through potential mechanisms of influence, enhancement of social networks and support. Implementation strategies will be developed in collaboration with partnering clinics and local Area Agencies on Aging. Participants will be recruited from three clinics at the University of Iowa Hospitals and Clinics (UIHC) that provide dementia diagnostic services and randomized into an intervention or control arm; and complete baseline and three- and six-month follow-up interviews. This study is innovative in its consideration of contributing factors at multiple levels of the ecological model (i.e., individual, social network, and organizational) and its collaborative approach, involving medical clinics, an Area Agency on Aging (AAA), and Alzheimer's Association (AA) to develop and evaluate a new care model that bridges between the medical and community settings.

DETAILED DESCRIPTION:
Once the participant has consented, the research assistant will set up a time to complete a baseline interview, either in-person or via telephone. The baseline interview will take 40-50 minutes to complete. After the baseline survey has been completed, the participant will be randomized using simple randomization based on a computer-generated random numbers to assign the family into the intervention or standard care (control group). If the participant is randomized into the intervention group, the options counselor will be given the participant's contact information and will establish contact with the participant to make an in-home or telephone (if preferred) visit within two weeks of the participant's consent. The participant and patient can jointly participate in the initial meeting. The options counselor may make additional calls to the participant if more information is needed in the absence of the patient as requested by the participant. During the initial visit/call, the options counselor will use the modified Options Counseling (OC) assessment tool and caregiver intake form (attached) to assess patient and family needs and to develop family actions plans (see attached family action plan form) using LifeLong Links to identify services available in their local areas, and to connect them to providers. The options counselor will also provide dementia education on the topics that the family desires to discuss. Modules to discuss with the participant include About Alzheimer's Disease and Dementia, Social Relationships and Daily Life, Anticipating Changes and Challenges, Interacting with Providers, and Addressing Future Needs. This initial visit should take between 1 and 2 hours. The options counselor will conduct 5 additional follow-up intervention calls, which will last between 30 minutes to 1 hour. These calls will happen each month, in the 5 months following the initial visit/call. The follow up intervention calls will be used to adjust action plans and implement additional training modules selected by the participant. The attached intervention log will be filled out by the options counselor after each session (6 sessions per participant) to track what was covered. The research team will use the intervention logs as fidelity checks. The sessions will also be recorded so that the research team can check for fidelity to intervention protocol. The options counselor, Maria Donohoe, is a research team member on this IRB.

Both intervention and standard care participants will complete 3 month and 6 month interviews, conducted by the research team members. The standard care group will have 3 and 6 month interviews prior to their receiving a call from an options counselor. The call and work that the standard care group does with an options counselor is not the intervention because the intervention protocol for this research will not be used. This phone call is made for the standard care group to receive support after the study data is collected if desired. Each follow up interview will take between 30 and 40 minutes to complete. All three interviews will be recorded so that research team members can review the data for accuracy. Participants will be asked by the research assistant for permission to record and will be invited to let the researcher know if they would not like to be recorded or if they would like to turn off the recorder at any time. Participants will still be able to participate in the study if they do not elect to be recorded. The responses questions will be recorded on paper and then entered into an online survey database on Qualtrics. Those in the intervention group wishing to continue and those in the standard care group wishing to receive Options Counseling after completing the 6 month interview will receive a call from a local options counselor in their area. Options Counseling services are provided using the Older American's Act funding by the local Area Agencies on Aging, thus, there will be no cost for older individuals and their family. . For each interview, the research assistant will make up to three calls to schedule a time, leaving a voicemail (if available) and a phone number to call if the participant would like to continue their participation. On the final call, the research assistant will let the participant know that this is the last call and if the participant would like to continue with the study, they are welcome to call back. Those who miss the 3-month follow-up interview will be contacted again for the 6-month follow up interview, and the same protocol will be used to establish contact.

At the end of the study (after the 6 month follow up interview), all study participants, regardless of study arm, will be given the option to receive a call from an options counselor who will offer options counseling services in their own community.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Speaks English
* Lives in Iowa
* Caregiver of someone diagnosed with dementia within the past 6 months

Exclusion Criteria:

- Does not meet inclusion criteria

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sato Ashida, PhD, Principal Investigator — University of Iowa; Kristine Williams, RN, PhD, Principal Investigator — University of Kansas
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rezende EL, Silva-Duran I I, Fernando Novoa F, Rosenmann M. Does thermal history affect metabolic plasticity?: a study in three Phyllotis species along an altitudinal gradient. J Therm Biol. 2001 Apr;26(2):103-108. doi: 10.1016/s0306-4565(00)00029-2. PMID 11163925
- [Derived] Ashida S, Lynn FB, Thompson L, Koehly LM, Williams KN, Donohoe MS. Using Clustering Methods to Map the Experience Profiles of Dementia Caregivers. Innov Aging. 2024 May 18;8(6):igae046. doi: 10.1093/geroni/igae046. eCollection 2024. PMID 38859822

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Options Counselor Health Educator Intervention Group | Control
Started | 42 | 40
Baseline interview | 42 | 40
3 month survey | 29 | 26
6 month survey | 25 | 25
Completed | 25 | 25
Not Completed | 17 | 15
Not completed — Lost to Follow-up | 12 | 14
Not completed — Death of care partner (person living with dementia) | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Options Counselor Health Educator Intervention Group | Control | Total
Number analyzed (Participants) | 42 | 40 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 31 | 28 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 16 | 11 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 41 | 37 | 78
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 41 | 37 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
FAST Score [Mean (Standard Deviation); unit: units on a scale] — Functional Assessment Staging Tool for dementia (FAST) is a measure of activity limitations due to dementia. The participant assessed their care partner (person living with dementia). The range is 1-7. A score of 1 is a normally functioning adult. A score of 7 is severe (end stages) of dementia.
  units on a scale | 2.5 (13.9) | 3.5 (13.3) | 3.0 (13.5)

OUTCOME MEASURES:

1. Primary Outcome: Modified Zarit Burden Interview
Description: Caregiver burden 12 item self report questionnaire; Minimum score 0, maximum score 36 with low scores showing less burden
Time Frame: Change over time from baseline to 6-month
Population: All participants who completed baseline. Note that the discrepancies in the number analyzed at different time points are due to patients dropping out of the study.
Measure: Mean (Standard Deviation); unit: Burden score
Groups:
- Options Counselor Health Educator Intervention Group: These individuals received the Options Counselor Health Educator (OC-HE) Intervention: The OC-HE met in person or over the telephone with the participant up to 6 times to provide options counseling based on modules developed by the research team.
- Control: These individuals received the typical standard of care treatment from clinics
Arm/Group | Options Counselor Health Educator Intervention Group | Control
Number analyzed (Participants) | 42 | 40
Burden score
  Baseline | 19.429 (9.399) | 17.950 (8.348)
  3-month: number analyzed (Participants) | 29 | 26
  3-month | 32.207 (7.466) | 27.160 (6.811)
  6-month: number analyzed (Participants) | 25 | 25
  6-month | 31.375 (6.864) | 28.615 (8.208)
Statistical Analysis 1: Comparison: Options Counselor Health Educator Intervention Group vs Control; Test type: Superiority; p = 0.206, Regression, Linear; We used generalized estimating equations to fit linear regression model for longitudinal data under the unstructured correlation matrix; Mean Difference (Net) = 1.128, Standard Error of Mean 1.622 — Estimated value: presented value is mean difference at month 6 from BL. Information from month 3 is included in the linear regression model. The reported p-value is the significance of the interaction effect between time and the intervention

2. Secondary Outcome: Knowledge of Formal Services
Description: Established measure of the extent to which caregiver knows about formal services available in their communities. Participants answer the extent to which (on a five-point Likert scale from "not at all true of me" to "completely true of me") they are informed about federal programs, that they know what to do to get help, that they know how to get the person they care for into a nursing home, that they are aware of how to pay for a nursing home, that they can get information about different options for getting care, that they know which home health care agencies are active in their area, that they know which nursing facilities are available in their area, and how to get assistance due to COVID (added later). The scale ranges from "Not True at all of me" to "Completely true of me", where these answers and those in between score 1-5. The scale is scored by adding up these scores of the 8 questions. Thus, the range is 8-40, with a 40 being the highest knowledge of formal services.
Time Frame: Change over time from baseline to 6-month
Population: Note that the discrepancies in the number analyzed at different time points are due to patients dropping out of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Options Counselor Health Educator Intervention Group | Control
Number analyzed (Participants) | 42 | 40
score on a scale
  Baseline | 25.381 (8.704) | 25.350 (8.678)
  3-month: number analyzed (Participants) | 29 | 26
  3-month | 29.690 (7.607) | 28.154 (7.953)
  6-month: number analyzed (Participants) | 25 | 25
  6-month | 29.520 (9.315) | 28.222 (7.567)
Statistical Analysis 1: Comparison: Options Counselor Health Educator Intervention Group vs Control; Test type: Superiority; p = 0.101, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.376, Standard Error of Mean 1.793 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Center for Epidemiologic Studies Depression
Description: Ten item measure assessing the extent to which the individual is experiencing depressive symptoms. Questions ask about how often feelings or events happen in a week on a scale from None of the time, where less than one day receives 0 points, to Most of the time, where 5 to 7 days receives 3 points. The lowest score is a 0, indicating no depression. The highest score is 30, indicating high depression.
Time Frame: Change over time from baseline to 6-month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Options Counselor Health Educator Intervention Group | Control
Number analyzed (Participants) | 39 | 36
score on a scale
  Baseline | 4.051 (4.751) | 2.806 (3.710)
  3-month: number analyzed (Participants) | 29 | 26
  3-month | 19.517 (7.740) | 19.640 (7.804)
  6-month: number analyzed (Participants) | 25 | 25
  6-month | 7.240 (6.741) | 5.815 (4.261)
Statistical Analysis 1: Comparison: Options Counselor Health Educator Intervention Group vs Control; Test type: Superiority; p = 0.836, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.201, Standard Error of Mean 1.174 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Emergency Care Use
Description: Self-reported measure of the number of times participants have visited a doctor or other health care provider unexpectedly in the past 6 months. The lowest score could be 0, indicating no emergency care use and the highest score for each could be 180 days, indicating that the participant visited a doctor or health care provider every day for the past six months
Time Frame: Change over time from baseline to 6-month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Options Counselor Health Educator Intervention Group | Control
Number analyzed (Participants) | 42 | 40
Visits
  Baseline | 0.714 (1.255) | 0.750 (1.296)
  3-months: number analyzed (Participants) | 29 | 26
  3-months | 0.207 (0.491) | 0.320 (0.476)
  6-months: number analyzed (Participants) | 25 | 25
  6-months | 0.292 (0.908) | 0.346 (0.562)
Statistical Analysis 1: Comparison: Options Counselor Health Educator Intervention Group vs Control; The outcome for this analyses is use of emergency care; Test type: Superiority; p = 0.567, Chi-squared; Mean Difference (Final Values) = 0.117, Standard Error of Mean 0.414 — Estimated value: presented value is for month 6. Since the outcome measure is count data, a log link function is used. The reported p-value is the significance of the interaction effect between time and intervention

5. Secondary Outcome: Social Network-Uplift
Description: Count of network members engaging in supportive interactions (Uplift) for each caregiver. Each caregiver had network members providing different levels of support. There are 8 survey questions to indicate whether network members engaged in uplifting interactions in any way. A network member with at least one interaction is counted. At each time point, the questions are asked again and reevaluated.
Time Frame: Change over time from baseline to 6-month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Count of support network members for a c
Arm/Group | Options Counselor Health Educator Intervention Group | Control
Number analyzed (Participants) | 41 | 40
Count of support network members for a c
  Baseline | 11.439 (6.786) | 10.750 (5.088)
  3-month: number analyzed (Participants) | 29 | 26
  3-month | 8.448 (5.494) | 12.400 (5.331)
  6-month: number analyzed (Participants) | 25 | 25
  6-month | 7.880 (5.102) | 9.889 (5.423)
Statistical Analysis 1: Comparison: Options Counselor Health Educator Intervention Group vs Control; Test type: Superiority; p = 0.014, Chi-squared; Mean Difference (Final Values) = -0.363, Standard Error of Mean 0.165 — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Social Network-Malfeasant
Description: Count of network members engaging in negative caregiving social interactions (Malfeasant) for each caregiver. Each caregiver had network members providing different levels of support. There are 7 survey questions to indicate whether network members engaged in malfeasant interactions in any way. A network member with at least one interaction is counted. At each time point, the questions are asked again and reevaluated.
Time Frame: Change over time from baseline to 6-month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Count of support network members for a c
Arm/Group | Options Counselor Health Educator Intervention Group | Control
Number analyzed (Participants) | 41 | 40
Count of support network members for a c
  Baseline | 2.098 (2.035) | 1.800 (1.436)
  3-month: number analyzed (Participants) | 29 | 26
  3-month | 4.966 (4.395) | 8.360 (5.992)
  6-month: number analyzed (Participants) | 25 | 25
  6-month | 1.520 (1.418) | 0.852 (1.027)
Statistical Analysis 1: Comparison: Options Counselor Health Educator Intervention Group vs Control; Test type: Superiority; p = 0.010, Chi-squared; Mean Difference (Final Values) = 0.467, Standard Error of Mean 0.301 — [estimate comment as in outcome 4, analysis 1]

7. Other Pre Specified Outcome: Caregiving Self-Efficacy
Description: 5-item self-reported measure assessing caregivers' confidence to use community-based services. The scale ranges on level of certainty from "not at all certain" to "very certain." The responses are scored on a scale of 0-10. These scores are summed up for a final score of 0-50, with a 50 being the highest knowledge of formal services. Questions include how certain the caregiver can get answers to all questions about services in the community, find organizations or agencies that provide services in need, arrange for services themselves, get answers to all questions about the individual's care, and get answers to changes in services due to the COVID-19 pandemic.
Time Frame: Change over time from baseline to 6-month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Options Counselor Health Educator Intervention Group | Control
Number analyzed (Participants) | 42 | 40
score on a scale
  Baseline | 29.524 (12.814) | 31.775 (10.666)
  3-month: number analyzed (Participants) | 29 | 26
  3-month | 35.345 (12.995) | 34.600 (10.528)
  6-month: number analyzed (Participants) | 25 | 25
  6-month | 33.667 (13.157) | 33.481 (7.992)
Statistical Analysis 1: Comparison: Options Counselor Health Educator Intervention Group vs Control; Test type: Superiority; p = 0.188, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 2.110, Standard Error of Mean 2.682 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 6 months
Description: No adverse events reported during this study. While some participants dropped the study due to a death, it was the death of the care partner (person living with dementia).
Groups:
- Options Counselor Health Educator Intervention Group: These individuals received the Options Counselor Health Educator Intervention
  Options Counselor Health Educator (OC-HE) Intervention: The OC-HE met in person or over the telephone with the participant up to 6 times to provide options counseling based on modules developed by the research team
Arm/Group | Options Counselor Health Educator Intervention Group | Control
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/40
Other Adverse Events (participants affected / at risk) | 0/42 | 0/40

LIMITATIONS AND CAVEATS:
This intervention trial was greatly affected by the COVID-19 pandemic resulting in small number of participants and modifications in recruitment and intervention delivery. Furthermore, it is hypothesized that this impact reduces power to detect the impact of the intervention. The impact of the pandemic was not accounted for in the statistical analyses while missing data may have occurred due to the pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT03932812/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT03932812/SAP_001.pdf
  • Informed Consent Form (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT03932812/ICF_002.pdf